CLINICAL TRIAL: NCT01054950
Title: Quality of Life in Food Allergic Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alan Baptist, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUM 33980
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and counseling (Experimental): Phone calls using behavioral techniques
  Interventions: Behavioral: Counseling
- Control (Placebo Comparator): Single phone call
  Interventions: Behavioral: Placebo phone call

INTERVENTIONS:
Behavioral: Counseling — Our food allergy nurse will contact our intervention group and discuss any questions or concerns they may have regarding their child's food allergy.
  Arms: Education and counseling
Behavioral: Placebo phone call — Phone call w/ no behavioral counseling
  Arms: Control

SUMMARY:
Food allergies are becoming more prevalent with more children being diagnosed with food allergies each year. Food allergies place a tremendous burden not just on the patient but on his/her family as well. In an attempt to provide better care to the investigators patients, the investigators would like to determine if regular contact with our food allergy nurse has a positive effect on a family's perceived quality of life.

DETAILED DESCRIPTION:
We intend to show a difference between the intervention group, who will receive a food allergy packet, along with three follow up phone calls from our trained allergy nurse, and the control group, will be given the food allergy packet only. We expect the intervention group to score higher on the quality of life survey, showing that the support and education of our allergy nurse has a positive effect on quality of life of our patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* IgE mediated food allergy
* Ages 0-17
* Willing to participate

Exclusion Criteria:

* Food sensitivities
* Unable to understand or read survey
* Unable to be available for follow up survey and nurse phone calls.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Difference in validated quality of life survey | twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, M.D, Study Director — University of Michigan Allergy and Immunology Clinic
Locations (1):
- University of Michigan Allergy and Immunology Clinic, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Baptist AP, Dever SI, Greenhawt MJ, Polmear-Swendris N, McMorris MS, Clark NM. A self-regulation intervention can improve quality of life for families with food allergy. J Allergy Clin Immunol. 2012 Jul;130(1):263-5.e6. doi: 10.1016/j.jaci.2012.03.029. Epub 2012 Apr 26. No abstract available. PMID 22541244